CLINICAL TRIAL: NCT05778942
Title: Multicentric Clinical Investigation on the Use of Preservative-Free Ophthalmic Solution Based on Sodium Hyaluronate and Xanthan Gum in the Treatment of Eye Discomfort, in Particular in Case of Ocular Dryness
Brief Title: Investigation of Preservative-Free Ophthalmic Solution in Ocular Dryness
Status: Completed | Type: Observational
Sponsor: SIFI SpA (Industry)
Responsible Party: Sponsor
Other Study IDs: 053/SI SYNFO
Record Dates: First submitted 2023-02-21; First posted 2023-03-22 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Dry Eye Syndromes
Keywords: Dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Arm: Single arm with commercial study drug: Eyestil SYNFO
  Interventions: Device: Eyestil SYNFO

INTERVENTIONS:
Device: Eyestil SYNFO — Instillation of study drug in both eyes: preservative-free ophthalmic solution based on sodium hyaluronate and xanthan gum

SUMMARY:
This is a multicenter, prospective, observational, open-label, non-interventional study evaluating the clinical performance and the safety of 4 daily instillations of the ophthalmic solution in the treatment of eye discomfort, in particular due to eye dryness

DETAILED DESCRIPTION:
Primary objective

▪ To evaluate the clinical performance of Eyestil SYNFO® as detected by the reduction of keratitis lesions objectified by corneal and conjunctival staining tests with fluorescein using the National Eye Institute (NEI) scale after 1 month of treatment compared to baseline.

Secondary objectives

* To evaluate the mean change of the corneal and conjunctival staining score with fluorescein using the NEI scale after 14 days of treatment and after 3 months of treatment compared to baseline.
* To evaluate conjunctival hyperemia index assessed by OCULUS Keratograph after 14 days, 1 month and 3 months of treatment compared to baseline.
* To evaluate the tear film stability as objectified by the tear film break-up time (TFBUT) test after 14 days, 1 month and 3 months of study treatment initiation compared to baseline.
* To evaluate the changes on the Best Corrected Visual Acuity (BCVA) measured by the "Early Treatment Diabetic Retinopathy Study" (ETDRS) after 14 days, 1 month and 3 months of study treatment initiation compared to baseline.
* To compare patients reported outcomes with baseline, using specifically:

  * the patient's reported Symptom Assessment questionnaire iN Dry Eye (SANDE) after 1 and 3 months of treatment;
  * the patient's Dry Eye-Related Quality-of-Life Score (DEQS) questionnaire after 1 and 3 months of treatment.
* To evaluate the safety and compliance of the medical device throughout the entire study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 years or older
* Subject able to provide Informed Consent, in compliance with Good Clinical Practice and local laws (thus, subject able to comprehend the full nature and purpose of the study, including possible risks and side effects)
* Subjects with ocular discomfort resulting from eye dryness in one or both eyes as determined by:

  * Scoring of ocular surface staining with fluorescein using the NEI scale (summing the score of cornea and conjunctiva, the total score per single eye range should be at least ≥6 on the 0-33 NEI scale)
  * TFBUT with fluorescein ≤10 seconds. The TFBUT value will be recorded as the average of 3 measurements
  * SANDE questionnaire ≥35
* Subject able to comply with the requirements of the clinical investigation plan, according to the Investigator

Exclusion Criteria:

* Corneal injuries or abrasions of traumatic origin
* Ocular infection or clinically significant inflammation (such as Herpes Simplex infection, corneal virus infection, bacterial, viral or fungal conjunctivitis, tuberculosis and mycosis of the eye, purulent and herpetic blepharitis, stye)
* Sjögren's syndrome
* Stevens-Johnson syndrome
* Concomitant treatment with drugs that may interfere with tear gland secretion
* Patients using any topical therapies such as non-steroidal anti-inflammatory drugs, cortisone, cyclosporine, vasoconstrictor, artificial tears (different than the investigated product)
* Treatment with topical or systemic corticosteroids in the 4 weeks preceding the study
* Known or potential hypersensitivity and/or history of allergic reactions to one of the components of the topical medical device
* Participation in another clinical trial within the previous 30 days
* Evidence of severe or uncontrolled systemic disease or any other significant disorders, which in the opinion of the Investigator does not allow the participation in the study or could compromise the results
* Pathologies associated with corneal thinning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects with signs and symptoms of ocular discomfort resulting from ocular dryness.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Keratitis lesions | 1 month
  To evaluate the clinical performance of Eyestil SYNFO® as detected by the reduction of keratitis lesions objectified by corneal and conjunctival staining tests with fluorescein using the National Eye Institute (NEI) scale after 1 month of treatment compared to baseline.

SECONDARY OUTCOMES:
Keratitis Lesions | Day 14 and at 3 months
  To evaluate the mean change of the corneal and conjunctival staining score with fluorescein using the National Eye Institute scale compared to baseline.
Conjuctival Hyperemia | Day 14, 1 month and 3 months
  To evaluate conjunctival hyperemia index by OCULUS keratograph
Best Corrected Visual Acuity | Day 14, 1 month and 3 months
  To evaluate changes in Best Corrected Visual Acuity (BCVA) using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score.
Tear Film Stability Break-Up time | Day 14, 1 month and 3 months
  The conjunctival tear film stability break-up time (TFBUT) will be evaluated after the instillation of 5 µl of a 2% preservative-free sodium fluorescein solution into the inferior conjunctival cul-de-sac- of each eye. The TFBUT value will be the average of 3 measurements.
SANDE Questionnaire | 1 and 3 months
  To compare patients reported outcomes with baseline, using the Symptom Assessment questionnaire iN Dry Eye (SANDE) questionnaire
DEQS Questionnaire | 1 and 3 months
  To compare patients reported outcomes with baseline, using the Dry Eye-Related Quality-of-Life Score (DEQS) questionnaire
Number of Adverse Events | From date of randomization up to 3 months
  To evaluate the safety through general assessment of adverse events
Investigator Global Assessment Score | From date of randomization up to 3 months
  To evaluate the safety using the Investigator Global Assessment Score
Intra Ocular Pressure | From date of randomization up to 3 months
  To evaluate the safety using the measurement of the intraocular pressure
Number and status (empty/unused) of returned devices | Day 14, 1 month and 3 months
  To evaluate compliance based on treatment administration and returned medical devices

CONTACTS AND LOCATIONS:
Overall Officials: Claudine Civiale, Study Director — SIFI S.p.A.
Locations (4):
- Spain (4):
  - Oftalvist, Alicante
  - Hospital Arruzafa, Córdoba
  - Hospital Clínico San Carlos, Madrid
  - Hospital Nuestra Señora de Gracia, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Molero Senosiain M, Burgos-Blasco B, Perez-Garcia P, Sanchez-Ventosa A, Villalba-Gonzalez M, Lopez Perez MD, Diaz JC, Diaz-Mesa V, Villarrubia Cuadrado A, Artiaga Elordi E, Larrosa Poves JM, Blasco A, Mateo A, Civiale C, Bonino L, Cano-Ortiz A. Performance and Safety of a Sodium Hyaluronate, Xanthan Gum, and Osmoprotectants Ophthalmic Solution in the Treatment of Dry Eye Disease: An Observational Clinical Investigation. Ophthalmol Ther. 2025 Apr;14(4):675-692. doi: 10.1007/s40123-025-01099-x. Epub 2025 Feb 21. PMID 39984804